CLINICAL TRIAL: NCT04446416
Title: An Open Label, Prospective, Pilot Study to Evaluate the Efficacy and Safety of Best Physician's Choice of Standard of Care Combined With NaviFUS System in Patients With Recurrent Glioblastoma Multiforme
Brief Title: Efficacy and Safety of NaviFUS System add-on Bevacizumab (BEV) in Recurrent GBM Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NaviFUS Corporation (Industry)
Collaborators: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NF-2019-01
Record Dates: First submitted 2020-06-16; First posted 2020-06-24 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Glioblastoma Multiforme; Glioblastoma; Glioma; Brain Tumor; Neoplasms; Neoplasms, Nerve Tissue
Keywords: NaviFUS System; Blood-Brain Barrier; Focused Ultrasound; GBM; Bevacizumab
MeSH Terms: conditions — Glioblastoma; Glioma; Brain Neoplasms; Neoplasms; Neoplasms, Nerve Tissue | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bevacizumab plus NaviFUS System (Experimental): Device: NaviFUS System BBB Disruption by FUS in recurrent GBM Microbubbles (MB) (SonoVue®) 0.1 mL/kg and optimal ultrasound exposure doses (based on the acoustic emission feedback FUS power control algorithm) generated from the NaviFUS System every 2 weeks to transiently open the BBB.
  Drug: Bevacizumab 10 mg/kg every 2 weeks for up to 36 weeks or until evidence of progressive disease, unacceptable toxicity, non-compliance with study follow-up, or withdrawal of consent.
  Interventions: Device: NaviFUS System; Drug: Bevacizumab

INTERVENTIONS:
Device: NaviFUS System — Open the BBB using focused ultrasound and contrast agent SonoVue®
Drug: Bevacizumab — An anti-angiogenic agent to block tumor growth
  Other Names: Avastin

SUMMARY:
This is a prospective, single-arm, two stages, open-label, pilot study to investigate the efficacy and safety of FUS add-on bevacizumab (BEV) in rGBM patients. The BEV is the best physician's choice of standard of care for rGBM after prior radiotherapy and temozolomide chemotherapy in the LinKou Chang Gung Memorial Hospital. Eligible patients will be enrolled through the process of informed consent.

DETAILED DESCRIPTION:
This trial will be divided into two stages. The study design and procedures will be as follows:

Stage 1:

Eligible patients will first be administered with BEV 10 mg/kg intravenous (IV) infusion. After 30-60 minutes, patients will receive microbubbles (MB) (SonoVue®) 0.1 mL/kg and optimal ultrasound exposure doses (based on the acoustic emission feedback FUS power control algorithm) generated from the NaviFUS System single exposure unit for up to two minutes every 2 weeks to transiently open the BBB.

After 4 weeks of treatment with BEV and single unit FUS-MB treatment, if the patient experienced BBB opening using FUS treatment and BEV IV infusion without any serious adverse effects (such as brain significant bleeding), then the patient may proceed to stage 2.

Stage 2:

Patients who complete stage 1 will enter stage 2 to receive the BEV with MB-mediated multiple units of FUS treatment for up to five minutes (but the maximum exposure time per single unit is two minutes) every 2 weeks for up to 30 weeks or until evidence of progressive disease, unacceptable toxicity, non-compliance with study follow-up, or withdrawal of consent.

After completion of study treatment, patients will be followed up for 28 days.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male/female patients ≥ 20 years of age
2. Patients with histologically confirmed glioblastoma, recurrent after prior radiotherapy and temozolomide chemotherapy.
3. Patient may have been operated for recurrence. If operated: with measurable residual tumor
4. Minimum interval since completion of radiation treatment is 12 weeks
5. Patients if already on the steroids then should be on a stable dose of steroids for at least 7 days prior to study treatment
6. Body mass index (BMI) ≥17 kg / m2
7. Minimum interval since last drug therapy:

   * 1 week for non-cytotoxic agents (e.g., interferon, tamoxifen), daily chemotherapy (e.g., metronomic temozolomide, cytoxan) or targeted therapies administered daily (e.g., gleevec, tarceva)
   * 4 weeks since last cytotoxic therapy
   * 6 weeks since the completion of a nitrosourea-containing chemotherapy regimen (e.g., carmustine (BCNU))
8. Patients with life expectancy ≥ 3 months
9. The Karnofsky performance status (KPS) in the patient must be > 60
10. Eastern Cooperative Oncology Group (ECOG) Score ≤ 2
11. Adequate hepatic, renal, coagulation, and hematopoietic function

    * Hemoglobin ≥ 8 g/dL
    * Platelets ≥ 100,000/mm3
    * Neutrophils ≥ 1,500/mm3
    * Serum creatinine ≤ 1.5 x upper limit of normal (ULN)
    * Urine protein creatinine (UPC) ratio < 1 or urine dipstick for proteinuria ≤ 2+
    * Alanine transaminase (ALT) < 3 ULN
    * Aspartate transaminase (AST) < 3 x ULN
    * Prothrombin time ≤ 1.2 x ULN
    * International Normalized Ratio (INR) < 1.5
    * Bilirubin < 2 x ULN
12. Patients with the region of interest (ROI) for FUS exposure are located close to the cortex with at least 20 mm distance beneath the skull bone and the ROI is not in the deep center brain with crucial brain functions, such as in the region of brain stem, or motor or speech regions
13. Patients with the potential for pregnancy and their partner must agree to use adequate contraception or be surgically sterile, or abstain from heterosexual activity starting with the first dose of treatment through at least 6 months after the last dose of BEV to avoid conception. Female patients of child-bearing potential must have a negative pregnancy test. Male patients must agree to use an adequate method of contraception starting with the first dose of treatment through 6 months after the last dose of BEV.
14. Able to give informed consent for the participation in the trial

Exclusion Criteria:

1. Patients who have had previous treatment with an inhibitor of vascular endothelial growth factor (VEGF) or VEGFR (including bevacizumab)
2. New York Heart Association (NYHA) Grade II or greater congestive heart failure requiring hospitalization within 12 months prior to screening
3. Severe hypertension at screening (diastolic blood pressure > 100 mmHg on medication)
4. Uncontrolled intercurrent illness including, but not limited to symptomatic congestive heart failure, unstable angina pectoris, severe cerebral or myocardial infarction, cardiac shunt, heart attack within the previous 12 months, stroke (except for transient ischemic attack; TIA) within the previous 6 months, or psychiatric illness/social situations that would limit compliance with study requirements
5. Unstable pulmonary disease or Chronic Obstructive Pulmonary Disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of screening
6. Implanted pacemaker, defibrillator or deep brain stimulator, other implanted electronic devices in the brain or documented clinically significant arrhythmias
7. Major surgery such as intra-thoracic, intra-abdominal or intra-pelvic (with the exception of craniotomy), open biopsy or significant traumatic injury ≤ 4 weeks prior to screening, or patients who have had minor procedures, percutaneous biopsies or placement of vascular access device ≤ 1 week prior to screening, or who have not recovered from side effects of such procedure or injury
8. Known HIV positive patients, however, that HIV testing is not required for entry into this study
9. Acute bacterial or fungal infection requiring intravenous antibiotics at the time of screening
10. Receiving anticoagulant (e.g. warfarin) or antiplatelet (e.g. aspirin) therapy within one week prior to beginning treatment
11. Pregnant or breast-feeding women
12. Known sensitivity/allergy to PET tracers, Magnetic Resonance Imaging (MRI) contrast agents, Computer Tomography (CT) contrast agents, SonoVue®, bevacizumab, or any of their components
13. Abnormal baseline findings considered by the investigator to indicate conditions that might affect study endpoints
14. Patients who have hemorrhage or cyst within the ROI
15. The receipt of an investigational drug within a period of 4 weeks prior to the first FUS exposure
16. Use of any recreational drugs or history of drug addiction
17. Any other condition that, in the investigator's judgment, might increase the risk to the patients or decrease the chance of obtaining satisfactory data needed to achieve the objectives of the study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-07-21 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2023-08-04 (Actual)

PRIMARY OUTCOMES:
Adverse Event | 38 weeks
  Number and severity of adverse event
Progression-free survival at 6 months (PFS-6) | 6 months
  Estimated rate of patients treated during 6 months without experiencing disease

SECONDARY OUTCOMES:
Tumor shrinkage | 38 weeks
  The tumor shrinkage rate (TSR) by measuring the longest diameter and perpendicular diameter of the main mass on MRI scans
Objective response rate (ORR) | 38 weeks
  Proportion of subjects in the analysis population who have complete response (CR) or partial response (PR) using Radiologic Assessment in Neuro-Oncology criteria (RANO) criteria
PET uptake | 38 weeks
  The uptake of PET (as standard uptake value - SUV and tumor-to-background ratio - TBR) in tumor and in normal contralateral gray matter before start of BEV+FUS treatment will be determined.
Overall survival (OS) | 38 weeks
  OS is defined as the time in months from study treatment to death or last follow-up if alive from any cause
Degree of the BBB opening | 38 weeks
  The FUS with microbubbles can temporally open the BBB. The spatial permeability of the BBB-opened region will be assessed using dynamic contrast-enhanced MRI (DCE-MRI).
Corticosteroid consumption | 38 weeks
  Increase or decrease in corticosteroid use compared to baseline. The mean corticosteroid dosage prior to study treatment will be considered as the patient's baseline.
Quality of life (QoL) assessment with the EORTC QLQ-C30 | 38 weeks
  The validated European Organization for Research and Treatment of Cancer (EORTC) quality of life questionnaire (QLQ-C30) will be used. The EORTC QLQ-C30 is a 30-item questionnaire. All of the response scale to questions are rated on a 4-point Likert scale from 1 = not at all, 2 = a little, 3 = quite a bit, to 4 = very much, and are linearly transformed to a 0-100 scale, with higher scores indicating more severe symptoms.
Quality of life (QoL) assessment with the EORTC QLQ-BN20 | 38 weeks
  The EORTC QLQ-BN20 is a QoL assessment specific to brain neoplasms. The questionnaire includes 20 items. All of the response scale to questions are rated on a 4-point Likert scale from 1 = not at all, 2 = a little, 3 = quite a bit, to 4 = very much, and are linearly transformed to a 0-100 scale, with higher scores indicating more severe symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Kuo-Chen Wei, M.D., Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Linkou Chang Gung Memorial Hospital, Taoyuan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liu HL, Hsu PH, Lin CY, Huang CW, Chai WY, Chu PC, Huang CY, Chen PY, Yang LY, Kuo JS, Wei KC. Focused Ultrasound Enhances Central Nervous System Delivery of Bevacizumab for Malignant Glioma Treatment. Radiology. 2016 Oct;281(1):99-108. doi: 10.1148/radiol.2016152444. Epub 2016 May 18. PMID 27192459
- [Background] Friedman HS, Prados MD, Wen PY, Mikkelsen T, Schiff D, Abrey LE, Yung WK, Paleologos N, Nicholas MK, Jensen R, Vredenburgh J, Huang J, Zheng M, Cloughesy T. Bevacizumab alone and in combination with irinotecan in recurrent glioblastoma. J Clin Oncol. 2009 Oct 1;27(28):4733-40. doi: 10.1200/JCO.2008.19.8721. Epub 2009 Aug 31. PMID 19720927
- [Background] Kreisl TN, Kim L, Moore K, Duic P, Royce C, Stroud I, Garren N, Mackey M, Butman JA, Camphausen K, Park J, Albert PS, Fine HA. Phase II trial of single-agent bevacizumab followed by bevacizumab plus irinotecan at tumor progression in recurrent glioblastoma. J Clin Oncol. 2009 Feb 10;27(5):740-5. doi: 10.1200/JCO.2008.16.3055. Epub 2008 Dec 29. PMID 19114704
- [Background] Mainprize T, Lipsman N, Huang Y, Meng Y, Bethune A, Ironside S, Heyn C, Alkins R, Trudeau M, Sahgal A, Perry J, Hynynen K. Blood-Brain Barrier Opening in Primary Brain Tumors with Non-invasive MR-Guided Focused Ultrasound: A Clinical Safety and Feasibility Study. Sci Rep. 2019 Jan 23;9(1):321. doi: 10.1038/s41598-018-36340-0. PMID 30674905
- [Background] Sonabend AM, Stupp R. Overcoming the Blood-Brain Barrier with an Implantable Ultrasound Device. Clin Cancer Res. 2019 Jul 1;25(13):3750-3752. doi: 10.1158/1078-0432.CCR-19-0932. Epub 2019 May 10. PMID 31076548
- [Derived] Chen KT, Tsai HC, Huang CY, Liau CT, Ho KC, Toh CH, Chuang CC, Hsu PW, Huang YC, Chang TW, Yeap MC, Chen PY, Lee CC, Lin YJ, Feng LY, Airan RD, Li G, Lim M, Liu HL, Wei KC. Combination of Neuronavigation-Guided Focused Ultrasound and Bevacizumab for Patients With Recurrent Glioblastoma: A Pilot Study. Neurosurgery. 2025 Nov 24. doi: 10.1227/neu.0000000000003851. Online ahead of print. PMID 41283685